CLINICAL TRIAL: NCT05139719
Title: A Phase IIb, Multi-center, Randomized, Double Blinded, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of HEC585 Tablets in Patients With Progressive Fibrosing Interstitial Lung Disease
Brief Title: A Study to Explore the Therapeutic Effect of HEC585 on Delaying Forced Vital Capacity (FVC) Decline and Tolerance in Progressive Fibrosing Interstitial Lung Disease (PF-ILD) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC585-PF-202
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Progressive Fibrosing Interstitial Lung Disease (PF-ILD) / Progressive Pulmonary Fibrosis (PPF)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HEC585 tables does A (Experimental)
  Interventions: Drug: HEC585 dose A
- HEC585 tables does B (Experimental)
  Interventions: Drug: HEC585 dose B
- placebo (Placebo Comparator): Placebo once daily up to 24 weeks in main stage; HEC585 dose A once daily up to 96 weeks in extended stage
  Interventions: Drug: HEC585 dose A; Drug: Placebo

INTERVENTIONS:
Drug: HEC585 dose A — taking HEC585 dose A orally once daily, up to 24 weeks in main stage (if applicable); up to 96 weeks in extended stage
  Arms: HEC585 tables does A; placebo
Drug: HEC585 dose B — taking HEC585 dose B orally once daily, up to 24 weeks in main stage; up to 96 weeks in extended stage
  Arms: HEC585 tables does B
Drug: Placebo — taking Placebo orally once daily, up to 24 weeks in main stage
  Arms: placebo

SUMMARY:
The main goal of this phase llb study is to compare the efficacy and safety of two doses of HEC585 tablets with placebo which is a look-alike substance that contains no active drug in patients with progressive fibrosing interstitial lung diseases. This study is divided into two stages, i.e. main study stage with 24 weeks treatment duration followed by up to 96 weeks treatment extended study stage.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the ICF.
2. Male or female patients' age ≥ 18 years when signing the ICF.
3. Patients with known or unknown etiology (except IPF) and clear pulmonary fibrosis on chest CT have undergone conventional clinical treatment (assessed by the investigator, including follow-up observation) for ≥ 3 months. At least two of the following criteria occurring within 12 months before screening without alternative explanation (such as infection, heart failure, etc.):

   i) Worsening respiratory symptoms like cough, shortness of breath. ii) Physiological evidence of disease progression (either of the following):
   1. absolute FVC (% of predicted) decline ≥ 5%.
   2. absolute DLco[Hb corrected] (% of predicted) decline ≥ 10%. iii) Radiological evidence of disease progression (one or more of the following):

   <!-- -->

   1. Increased extent or severity of traction bronchiectasis and bronchiolectasis.
   2. New ground-glass opacity with traction bronchiectasis.
   3. New fine reticulation.
   4. Increased extent or increased coarseness of reticular abnormality.
   5. New or increased honeycombing.
   6. Increased lobar volume loss.
4. Fibrosing lung disease on HRCT, defined as reticular abnormality with traction bronchiectasis with or without honeycombing, with disease extent of >10% as confirmed by central readers.
5. For patients with underlying connective tissue disease (CTD) should be in the stable status which is defined by no initiation of new therapy, treatment dose adjustment or withdrawal of therapy within 12 weeks prior to randomization.
6. FEV1/FVC ≥ 0.7 before using bronchodilators.
7. %FVC ≥ 45% predicted.
8. Carbon Monoxide Diffusion Capacity (DLCO) corrected for Haemoglobin (Hb) ≥ 30% and ≤ 80% predicted of normal.
9. Fertile female or male subjects agreed and promised to take effective contraception measures from signing the ICF till 30 days after last administration.
10. Subjects are willing and able to comply with the protocol requirements and attend visits assessed by the investigator.

Exclusion Criteria:

1. Diagnosis of Idiopathic Pulmonary Fibrosis (IPF).
2. Lung with other clinically significant abnormalities which the investigator assess to have an effect on the results of study.
3. Significant Pulmonary Arterial Hypertension (PAH), such as meeting the following: Previous clinical or echocardiographic evidence of significant right heart failure, History of right heart catheterization showing a cardiac index ≤ 2 L/min/m², or PAH requiring parenteral therapy with epoprostenol/treprostinil.
4. Major extrapulmonary physiological or pathological restriction (e.g. chest wall abnormality, large pleural effusion).
5. Expected to receive lung transplantation during the study.
6. Expected survival time is less than 6 months.
7. History of malignant tumors within 5 years (except for localized cancers such as basal cell carcinoma and carcinoma in situ of cervix).
8. Thyroid dysfunction that the investigator assessed to be clinically significant and needed to be treated.
9. History of unstable or worsening heart disease during the 6 months prior to screening, including but not limited to the following:

   1. Unstable cardiac angina,
   2. Acute Myocardial infarction,
   3. Congestive heart failure (need to be treated in hospital or NYHA III/IV),
   4. Uncontrolled Severe Arrhythmias.
10. TBIL >1.2 × ULN, AST or ALT > 1.5 × ULN.
11. CLcr < 50 mL/min.
12. Human immunodeficiency virus (HIV) or treponema pallidum antibody is positive.
13. Uncontrolled hepatitis B virus infection or hepatitis C virus infection.
14. Use of any of the following medications for the treatment of Interstitial Lung Disease (ILD) or influence the effect or safety of investigational drug:

    1. Strong inducers or strong inhibitors of CYP3A4 within 4 weeks before randomization.
    2. Azathioprine (AZA), cyclosporine, MMF ( > 1.5 g/d or equivalent dose), tripterygium glycosides , hydroxychloroquine, tacrolimus, prednisone > 15mg/day or equivalent systemic glucocorticoid therapy, and the combination of OCS+AZA+NAC within 4 weeks before randomization.
    3. Cyclophosphamide within 8 weeks before randomization.
    4. Combination of ≤ 15mg/day or equivalent systemic glucocorticoid therapy with ≤ 1.5 g/d or equivalent dose MMF within 12 weeks before randomization.
    5. Pirfenidone or nintedanib within 1 months before screening.
    6. Rituximab, Adalimumab, Secukinumab, Infliximab, Tocilizumab, Certolizumab, Golimumab, Tofacitinib, Baricitinib, Etanercept, Abatacept within 6 months before randomization.
15. Subjects cannot complete the PFT、6MWT,or questionnaires.
16. Allergic to any component of HEC585 Tablets.
17. Participated in other clinical study and received the last dose within 3 months before screening.
18. Pregnant or breastfeeding.
19. History of smoking (≥ 10 cigarettes/day) within 3 months before screening or are unwilling to quit smoking during the study.
20. History of alcohol or drug abuse within 6 months before the screening.
21. Any condition that, in the opinion of the investigator, would compromise the safety or compliance of the subject, or prevent the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 24 in FVC (mL) compared with placebo | 24 Weeks
  change in FVC (mL), measured using Spirometer, from baseline to week 24

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in FVC (mL) compared with placebo | 12 Weeks
  change in FVC (mL), measured using Spirometer, from baseline to week 12
Proportion of subjects with the decline from baseline in FVC (% predicted) > 10% | 24 Weeks
  The proportion of subjects whose %FVC decline from baseline by more than 10% in each treatment group at week 24
Proportion of subjects with the decline from baseline in FVC (% predicted) > 5% | 24 Weeks
  The proportion of subjects whose %FVC decline from baseline by more than 5% in each treatment group at week 24
Changes of DLco (Hb correction) | 12 Weeks, 24 Weeks
Changes of 6MWT results | 12 Weeks, 24 Weeks
Changes of St George' s Respiratory Questionnaire (SGRQ) | 12 Weeks, 24 Weeks
  The higher the score, the more serious the impact on life
Changes of The University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) | 12 Weeks, 24 Weeks
  Scores range from 0 to 120. The higher the score, the more severe the difficulty in breathing
Changes of Leicester coughing questionnaire scores | 12 Weeks, 24 Weeks
  Scores range from 3 to 21. The lower the score, the greater the impact of cough on quality of life
Changes of HRCT | 24 Weeks
Time to first acute ILD exacerbation or death | 24 Weeks
  the time duration from randomization to first acute ILD exacerbation or death whichever occurs first
Proportion of subjects with death caused by any reason(s) | 24 Weeks
Proportion of subjects with death caused by the respiratory reason | 24 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No